CLINICAL TRIAL: NCT03098485
Title: Prospective Study Characterizing Fecal Microbiome Disruptions During and After Receipt of Antimicrobials
Brief Title: Healthy Patients & Effect of Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201610071
Record Dates: First submitted 2017-01-11; First posted 2017-03-31 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Microbiota; Anti-bacterial Agents
MeSH Terms: interventions — Levofloxacin; Ofloxacin; Azithromycin; Cefpodoxime; Cefpodoxime Proxetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Levofloxacin (Experimental): 1 750mg tab of levofloxacin by mouth for 5 days
  Interventions: Drug: Levofloxacin
- Azithromycin (Experimental): 1 500mg tab by mouth on day 1, then 1 250 mg tab per day by mouth for 4 days (total 5 days)
  Interventions: Drug: Azithromycin
- Cefpodoxime (Experimental): 200mg tab by mouth twice per day for 5 days
  Interventions: Drug: Cefpodoxime
- Azithromycin and cefpodoxime (Experimental): Azithromycin: 1 500mg tab by mouth on day 1, then 1 250 mg tab per day by mouth for 4 days (total 5 days)
  Cefpodoxime: 200mg tab by mouth twice per day for 5 days
  Interventions: Drug: Azithromycin; Drug: Cefpodoxime

INTERVENTIONS:
Drug: Levofloxacin — 5 days of levofloxacin administration
  Other Names: Levaquin, Quixin, Iquix
  Arms: Levofloxacin
Drug: Azithromycin — 5 days of azithromycin administration
  Other Names: Zithromax, AzaSite, Zmax
  Arms: Azithromycin; Azithromycin and cefpodoxime
Drug: Cefpodoxime — 5 days of cefpodoxime administration
  Other Names: Vantin
  Arms: Azithromycin and cefpodoxime; Cefpodoxime

SUMMARY:
The objective of this study is to evaluate the impact of antimicrobial (antibiotic) exposures on the microbiome in healthy adults, specifically during and after usual courses of the antimicrobials used to treat community acquired pneumonia (CAP). Pneumonia is a lung infection, and community-acquired pneumonia is pneumonia that develops outside of a healthcare facility (i.e., in the community). A microbiome is a the community of microorganisms living in a particular location, such as the gut or the mouth. Disruptions to a person's microbiome may reduce his/her "colonization resistance" (resistance to colonization with pathogenic microorganisms) and make him/her more susceptible to multidrug resistant organism (MDRO) colonization and infection.

To study changes in the microbiome, the investigators will recruit 20 healthy adult volunteers and obtain fecal, salivary, skin, and urine specimens at multiple time points before, during, and after administration of antimicrobials. Participants will be randomized to one of 4 antimicrobial regimens, all of which are FDA-approved for treatment of community-acquired pneumonia. Stool specimens will be analyzed via stool culture and genetic sequencing, and all remaining specimens will be frozen and used to create a biospecimen repository for future analysis. The rationale for using healthy volunteers (instead of patients already prescribed antibiotics by their physicians) is because the human microbiome is very complex and can be affected by a variety of medical conditions and other medications. In addition, the presence or absence of patient-specific factors means people with infections may not be prescribed the specific courses of antibiotics the investigators are trying to study. Studying the effect of antibiotics on healthy volunteers will provide baseline data that are more applicable to the population at large.

DETAILED DESCRIPTION:
Each year, antimicrobial resistance causes over two million infections and 23,000 deaths in the US alone, representing a critical global public health issue. Some of the most feared multidrug resistant organisms (MDROs) include Clostridium difficile, carbapenem-resistant Enterobacteriaceae (CRE), extended spectrum beta-lactamase producing Enterobacteriaceae (ESBL), MDRO Acinetobacter, and MDRO Pseudomonas aeruginosa; there are few antimicrobials effective against these MDROs, and available antimicrobials often have rate-limiting toxicities. The major risk factor for MDRO colonization and subsequent MDRO infections is exposure to antimicrobials. The use of antimicrobials has been associated with an altered and often less diverse composition of the fecal microbiome, and expansion of the resistome. A "healthy" microbiome provides "colonization resistance" against potentially pathogenic bacteria; antimicrobials disrupt this protective community, providing selective pressure that favors MDRO colonization, persistence, and transmission to others.

Methods to proactively prevent MDRO colonization, rather than reliance on reactive approaches to this problem, are urgently needed. Antimicrobial stewardship is a key component of MDRO prevention efforts; however, there is no method to determine which antimicrobials cause the greatest degree of microbiome disruption. A better understanding of exactly how antimicrobials alter the microbiome is necessary to optimally guide future MDRO prevention efforts and antimicrobial stewardship. The development of microbiome disruption indices (MDIs) would help characterize the risk associated with specific antimicrobials, and can be used during antimicrobial development, patient monitoring while on antimicrobials, and to facilitate infection prevention efforts to contain MDRO spread. Additionally, MDIs can be used as an alert when microbiome disruptions reach a critical level and MDRO colonization is imminent. At that point, interventions to restore the microbiome could be implemented.

Community-acquired pneumonia (CAP) is one of the leading causes of death in the United States, with an estimated >900,000 cases each year in adults age 65 and older. Large amounts of antimicrobials are used in treating patients with CAP because the disease is relatively common. A better understanding of the effect of CAP antimicrobial treatment on the microbiome could result in improved treatment options for patients with CAP and protect CAP patients from colonization or infection with MDROs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 21-60 residing in the St. Louis, Missouri, USA metropolitan area

Exclusion Criteria:

* History of allergic reaction to study antimicrobial(s)
* Contraindication(s) to study antimicrobial(s)
* Inability to provide regular stool samples
* Any non-topical antimicrobial exposure in previous 6 months
* Tube feeds as primary source of nutrition in previous 6 months
* Pregnant or risk of becoming pregnant during study period
* Breastfeeding during study period
* Gastroenteritis in last 3 months
* Any non-elective hospitalization in the previous 12 months
* Incontinent of stool
* Known colonization with an MDRO
* Anticipated change in diet or medications during study period
* Elective surgery during study period
* History of an intestinal disorder
* Inability to provide written, informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01; Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennie H. Kwon, DO, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Summarized metagenomics sequence data will be made available through public repositories at the time of manuscript publication.

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin and Cefpodoxime: Azithromycin: 1 500mg tab by mouth on day 1, then 1 250 mg tab per day by mouth for 4 days (total 5 days)
  Cefpodoxime: 200mg tab by mouth twice per day for 5 days
  Azithromycin: 5 days of azithromycin administration
  Cefpodoxime: 5 days of cefpodoxime administration
Period: Overall Study
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Customized [Median (Full Range); unit: years]
  Age (years) | 41 [40 to 59] | 27 [26 to 41] | 39 [24 to 53] | 34 [26 to 37] | 37 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 2 | 10
  Male | 3 | 4 | 0 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 4 | 4 | 5 | 4 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Degree of Microbial Disruption: Number of Patients With Recovery of Bacterial Species Richness at 185 Days Post-antibiotics
Description: The degree of microbial disruption will be defined by recovery of bacterial species richness (number of species) after antibiotics.
Time Frame: Decrease from baseline (7 days prior to antibiotics) in microbial diversity at 185 days post-antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 3 | 3 | 2 | 3

2. Primary Outcome: Degree of Microbial Disruption: Number of Patients With Increase in Antibiotic Resistance Genes at 185 Days Post-antibiotics
Description: The degree of microbiome disruptions will be defined by an increase in the number of antibiotic resistance genes after antibiotics compared to baseline.
Time Frame: Increase from baseline (7 days prior to antibiotics) in antibiotic resistance genes at 185 days post-antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 4 | 5 | 5 | 4

3. Primary Outcome: Degree of Microbial Disruption: Number of Patients With Continued Microbial Disruption at 185 Days Post-antibiotics
Description: The degree of microbiome disruptions will be defined by continuing microbial disruption, as measured by Bray-Curtis dissimilarity, post-antibiotics compared to baseline.
Time Frame: Persistent disruption from baseline (7 days prior to antibiotics) in microbial composition at 185 days post-antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants | 4 | 4 | 5 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Levofloxacin | Azithromycin | Cefpodoxime | Azithromycin and Cefpodoxime
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03098485/Prot_SAP_000.pdf